CLINICAL TRIAL: NCT01757548
Title: The Effect and Prognosis of Different Operations on Varicocele - a Single-center Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Bing Yao, graduate student, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2011010005282
Record Dates: First submitted 2012-12-14; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Varicocele; Male Infertile;Varicocelectomy
Keywords: varicocele; male infertile;varicocelectomy
MeSH Terms: conditions — Varicocele | interventions — Microsurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- open operation (Experimental): high ligation of spermatic vein by open operation
  Interventions: Procedure: open operation
- microsurgery (Experimental): high ligation of spermatic vein by microsurgery
  Interventions: Procedure: microsurgery

INTERVENTIONS:
Procedure: open operation — high ligation of spermatic vein by open operation
  Arms: open operation
Procedure: microsurgery — high ligation of spermatic vein by microsurgery
  Arms: microsurgery

SUMMARY:
The purpose of this study is to determine whether high ligation of spermatic vein by open operation and microsurgery for patients with are effective in the treatment of varicocele and to determine which surgical option is better.

ELIGIBILITY:
Inclusion Criteria:

* 1.infertile patient suffering from varicocele 2.severe varicocele patient with obvious symptoms 3.adolescents suffering from severe varicocele with or without orchiatrophy

Exclusion Criteria:

* 1.varicocele patient with abdominal infection 2.varicocele patient who has massive adhesion of pelvic tissue due to pelvic surgery history 3.mild varicocele 4.varicocele patient has no obvious symptoms if has have born children, suffer from idiopathic azoospermia，or their partner can't bear children

Ages: 10 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
the quality of semen and the level of sexual hormone | before and three and six months after surgery
  The semen analyses and were sexual hormones determinations conducted before and three and six months after surgery.Then the quality of semen and the level of sexual hormone before and after surgery were compared.
complications | one, three and six months postoperation
  the complications such as recurrence, hydrocele,orchiatrophy and wound infection were assessed one, three and six months postoperation. Color doppler ultrasonography and physical examination are the main methods to assess the complications

SECONDARY OUTCOMES:
If there was pain, visual analogue scale,Numerical rating scale and verbal rating scale would be used to evaluate pain intensity. pain intensity | before and one,three and six months after surgery
  If there was pain, visual analogue scale,Numerical rating scale and verbal rating scale would be used to evaluate pain intensity.

OTHER OUTCOMES:
general information | before surgery
  Before surgery, all patients were diagnosed by physical examination and testified by color Doppler ultrasound. And we documented the patients' age, left unilateral or bilateral and the grade of varicocele

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Zhou Sun, MD，PhD, Study Director — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- First Affiliated hospital，Sun Yat-Sen University., Guangzhou, Guangdong, China